CLINICAL TRIAL: NCT03738254
Title: Motivating Survey Compliance: Game Play Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1708061907
Record Dates: First submitted 2018-11-07; First posted 2018-11-13 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Patient Reported Outcome Measures; Compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Paper PRO (Active Comparator): Participants in the Paper PRO arm completed daily patient reported outcome diaries on paper
  Interventions: Other: Paper Survey
- ePRO (Active Comparator): Participants in the ePRO arm completed daily patient reported outcome diaries online via a smartphone app.
  Interventions: Other: Electronic Survey
- Game-Motivated ePRO (Experimental): Participants in the Game-Motivated ePRO arm completed daily patient reported outcome diaries online via a smartphone app. These participants were also given access to a game that rewarded the participant with an in-game reward that helped the participant complete various in-game quests.
  Interventions: Other: The Guardians: A smartphone game

INTERVENTIONS:
Other: The Guardians: A smartphone game — "The Guardians" is a mix of two popular game genres: idle games (a game that doesn't require constant player input in order to progress in the game, but often progresses exponentially in response to a few user inputs, e.g., Cookie Clicker and Adventure Capitalist) and pet collection games (a game where the player seeks to collect all of the pets in a set, e.g., Pokemon or Neko Atsume). The game gives the player an in-game reward for completing a survey.
  Arms: Game-Motivated ePRO
Other: Paper Survey — Paper version of daily survey
  Arms: Paper PRO
Other: Electronic Survey — Electronic version of daily survey administered via a smartphone app.
  Arms: ePRO

SUMMARY:
Self-reports, especially for patients with chronic physical or mental diseases, are critical for disease research and drug development. Historically, it has been very difficult to collect self-reported data for long periods of time as it is an unpleasant and inconvenient task. Paper and digital surveys are the traditional way of collecting self-reports and have been around for a long time, but still suffer from lack of adherence despite the best efforts of researchers to remind and motivate individuals to fill them out.

Mobile games, on the other hand, benefit from an enormous amount of human adherence. These video games can be played on a smartphone and have captured the attention of a wide variety of demographics. The investigators have used established game design principles to develop a mobile game to motivate individuals to fill out a daily survey.

The purpose of this study is to determine which method of survey administration (paper, digital survey, or game- motivated survey) leads to the highest adherence rates for daily surveys.

DETAILED DESCRIPTION:
The recruitment flyers, emails, and postings will invite eligible individuals to participate in a 35-day study about mood, games, and time use for $100. Interested persons will be invited to go to a link to fill out a screening survey. Potential participants will be screened to make sure they are in the appropriate age range and have a smartphone. This will be accomplished via an online survey.

Once a potential participant has been identified, he or she will be directed to digital information about the study that is written in an easily understandable format. This information will include the types of questions that will be asked on a daily basis, information about the pre- and post- surveys, information about payment ($40 for finishing the first 4 of 7 surveys and an additional $60 for finishing the post-study survey), and notification that the participant does not need to fill out any question if it makes him/her uncomfortable. If the individual still wants to participate, they will be instructed to enter the email address of a parent or guardian who can provide consent for them. If the individual is 18 years old or older, they will provide their own consent. Individuals under 18 will read and digitally sign an assent form.

After a participant has consented to participate, he or she will be randomized into one of 3 groups for filling out the daily surveys: paper surveys, digital surveys, or game-motivated digital surveys. The participant will then fill out a pre-study survey about general demographics (age, gender), gaming and time use habits, and complete a couple of quick assessments to determine reading level and arithmetic level. Then participants will provide an email address to receive payment at the end of the study. Participants will be reminded of the payment schedule and then be directed to download the free app that matches his or her randomized group. Note that the paper surveys group will visit a webpage that displays a randomized word that he or she will need to write on the paper survey so that we can approximate when the survey was filled out. In addition, the paper surveys group participants will also be directed to print out their surveys for the study.

After the pre-study survey is complete, participants will receive a daily notification from their downloaded app to remember to fill out their survey for the day for 35 days. Each participant will be asked the following 5 questions each day:

1. What was your mood during the last 24 hours?
2. How many minutes did you spend playing mobile games in the last 24 hours?
3. How many times did you watch ads for in-game rewards in the past 24 hours?
4. How many minutes did you spend outside in the last 24 hours?
5. What has the weather been like in the last 24 hours?

Additionally, participants in the paper survey will be required to write the word that is on the webpage. This allows us to get an approximation of when the paper survey was filled out.

In the digital survey, we will record the time taken to complete each question and the latency between the notification to complete the survey and the actual survey completion. In the game-motivated survey, we will also record the participant's interactions with the game.

Once the 35-day study is over, participants will be sent a link to fill out the post-study survey. Participants in the paper survey group will also be given instructions for returning the forms to us via FedEx (participants will be given $10 to cover any charges incurred for returning the surveys).

Participants will then be sent their compensation in the form they indicated (Amazon Giftcard via email).

Analysis will be completed to compare average completion rates between the three study arms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-24
* Own and use either an iPhone or Android smartphone
* Access to US Apple App Store or US GooglePlayStore

Exclusion Criteria:

* N/A

Ages: 6 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 232 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
Adherence Rates to various methods of daily survey administration | 35 days
  For each study arm, the average adherence rate (computed as the percent of days (out of 35 total) a participant completed 100% of the daily survey questions, averaged over all participants in the study arm) will be computed and compared

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind W Picard, ScD, Principal Investigator — Massachusetts Institute of Technology
Locations (1):
- Massachusetts Institute of Technology, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taylor S, Ferguson C, Peng F, Schoeneich M, Picard RW. Use of In-Game Rewards to Motivate Daily Self-Report Compliance: Randomized Controlled Trial. J Med Internet Res. 2019 Jan 3;21(1):e11683. doi: 10.2196/11683. PMID 30609986